CLINICAL TRIAL: NCT01305174
Title: Balloon Expandable vs. Selfexpanding Stents to Treat Stenosis or Occlusions of Common and External Iliac Artery Disease
Brief Title: Iliac, Common and External (ICE) Artery Stent Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Delayed recruitment
Sponsor: Medical Care Center Prof. Mathey, Prof. Schofer, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICE 3.0
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Vascular Lesions
Keywords: Common Iliac Artery and External Iliac Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balloon expandable stent arm (Active Comparator): First placement of the sheath and successful passage of a 0.018" or 0.035" guidewire via the sheath across the target lesion in the iliac arteries was required. Consecutively the balloon-expandable stent (Visi-Pro™, ev3 Endovascular, Inc., Plymouth, MN, USA), which was premounted on a balloon catheter, was deployed by inflation of the balloon. The nominal stent diameter had to approximate the reference vessel diameter of the target lesion. Postdilation was permitted
  Interventions: Device: PROTEGE GPS stent vs. VISI-PRO stent
- Selfexpanding stent arm (Active Comparator): First placement of the sheath and successful passage of a 0.018" or 0.035" guidewire via the sheath across the target lesion in the iliac arteries was required. Consecutively the the self-expanding stent (Protege™, ev3 Endovascular, Inc., Plymouth, MN, USA), which had to exceed in the nominal diameter the reference vessel diameter at least by 1 mm, was released. Postdilation was mandatory. The inflated postdilation-balloon should approximate the reference vessel diameter.
  Interventions: Device: PROTEGE GPS stent vs. VISI-PRO stent

INTERVENTIONS:
Device: PROTEGE GPS stent vs. VISI-PRO stent — Visi-Pro balloon expandable stent vs. PROTEGE GPS selfexpanding nitinol stent to treat stenosis or occlusion of common and external iliac artery disease
  Other Names: ev3; peripheral stents; iliac artery; PAOD

SUMMARY:
The objective of this prospective, randomized,controlled and multicenter trial is, to compare recurrent-restenosis rates in the balloon expandable VISIO-PRO stent arm and the selfexpandable PROTEGE GPS stent arm 12 month after treatment of stenosis or occlusions of common and external iliac artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years.
2. Patient must sign informed consent form.
3. Patient must agree to participate in the study and comply with follow-up requirements.
4. Clinically, all patients must be in Rutherford category 1 to 4.

   Angiographic Inclusion Criteria:
5. Planned stenting (degree of stenosis 70-100%) within the common or external iliac artery. The target lesion must not extend beyond the iliac arteries.
6. Lesion segment starts at the aortic bifurcation and ends at the take off of the common femoral artery (Offset of the iliac circumflex artery beneath the ligamentum inguinale).
7. The length of the lesion should be at least 1 cm and maximally 20 cm (measurement by radiopaque ruler).
8. The degree of target lesion stenosis must be determined by pre-interventional duplex ultrasound or (MR-) angiography.
9. Patency of ipsilateral profunda artery. Ipsi- or contralateral artery lesions of the leg can be treated prior to the treatment of the study lesion.
10. In cases of two or more stenotic regions within the segment, these are considered separate lesions if there is a nonstenotic or only mildly stenotic (< 30%) segment of at least 2 cm in length between them. Otherwise, they are considered as single lesion. In case of separate lesions, only the proximal lesion will be taken as the target lesion!
11. A tandem lesion that can be treated with one stent will be considered as one lesion.

Exclusion Criteria:

1. Patient is currently participating in another clinical trial
2. Pregnancy or pregnancy planned during study duration
3. Life expectancy less than 2 years
4. Co-morbidities preventing study participation
5. Severe coagulation disorders
6. Current treatment with anticoagulants other than aspirin, ticlopidine, clopidogrel or prasugrel.
7. Active gastric ulcer or gastrointestinal bleeding
8. Thrombotic occlusion of the target vessel within previous 4 weeks.
9. Treatment of target lesion with laser or atherectomy devices.
10. Dialysis dependency.
11. Manifest hyperthyreosis.
12. Known allergy against contrast agent that cannot be adequately controlled by usual premedication.
13. Known heparin intolerance.
14. Known paclitaxel intolerance.

    Angiographic:
15. Target lesion extends into the femoral artery.
16. Symptomatic untreated inflow lesion > 70% in ipsilateral iliac arteries. Pretreatment of iliac stenosis is possible.
17. Target Lesion is in aortic bifurcation and needs treatment with "kissing balloon technique"
18. Lesion in abdominal aorta that needs treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Duplex-ultrasound determined recurrent restenosis after 12 month | 12 month
  Duplex-ultrasound definition:
  = recurrent stenosis ≥ 70% in relation to vessel diameter or PSV >3.4 per duplex ultrasound

SECONDARY OUTCOMES:
Clinical improvement of walking distance and improvement of at least 1 Rutherford category | 12 and 24 month
  Clinical improvement of walking distance and improvement of at least 1 Rutherford category
Improvement of ABI of at least o.1 points in treated leg after 6 and 12 month (AHA Guidlines) | 6 and 12 month
Clinically driven target lesion revascularization (TLR and TVR) at 6 and 12 month | at 6 and 12 month
  TLR = Target Lesion Revascularisation TVR = Target Vessel Revascularisation
Recurrent stenosis >= 70%within the stent at 6 and 12 month | at 6 and 12 month
Clinical and hemodynamic parameters (walking distance, ABI, Rutherford category) at 1, 6 and 12 month | at 1, 6 and 12 month
Primary angiographic success rate (<30% residual stenosis) | Procedure
Major adverse vascular events plus death rate | 24 month
  Major adverse vascular events plus death rate

CONTACTS AND LOCATIONS:
Overall Officials: Hans Krankenberg, Dr., Principal Investigator — Medical Care Center Prof. Mathey, Prof. Schofer
Locations (1):
- Medical Care Center Prof. Mathey, Prof. Schofer, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Krankenberg H, Zeller T, Ingwersen M, Schmalstieg J, Gissler HM, Nikol S, Baumgartner I, Diehm N, Nickling E, Muller-Hulsbeck S, Schmiedel R, Torsello G, Hochholzer W, Stelzner C, Brechtel K, Ito W, Kickuth R, Blessing E, Thieme M, Nakonieczny J, Nolte T, Gareis R, Boden H, Sixt S. Self-Expanding Versus Balloon-Expandable Stents for Iliac Artery Occlusive Disease: The Randomized ICE Trial. JACC Cardiovasc Interv. 2017 Aug 28;10(16):1694-1704. doi: 10.1016/j.jcin.2017.05.015. PMID 28838480
- See also: Study website in german — http://www.icetrial.de